CLINICAL TRIAL: NCT06833567
Title: Brief Mentalization-based Group Psychotherapy for Anxiety and Depression Disorders and Spanish Cultural Adaptation and Validation of the Epistemic Trust Questionnaire (QET)
Brief Title: Mentalizing and Epistemic Trust in Patients With Anxiety and Depression.
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Fundación Pública Andaluza para la Investigación de Málaga en Biomedicina y Salud (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MENT/CE_24
Record Dates: First submitted 2025-02-13; First posted 2025-02-18 (Actual); Last update posted 2025-02-18 (Actual); Status verified 2025-02

CONDITIONS: Anxiety Disorders; Depression
MeSH Terms: conditions — Anxiety Disorders; Depression

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Brief mentalization-based group psychotherapy (Experimental): Participants will attend mentalization-based psychotherapy group sessions of 12 weekly sessions.
  Interventions: Behavioral: Brief mentalization-based group psychotherapy
- Acceptance and commitment therapy group intervention (Active Comparator): Participants will attend to usual group intervention based on Acceptance and Commitment Therapy of 12 weekly sessions.
  Interventions: Behavioral: Acceptance and Commitment Therapy group intervention

INTERVENTIONS:
Behavioral: Brief mentalization-based group psychotherapy — The intervention is an adaptation for anxiety and depression profiles of the introductory group program to Mentalization-Based Treatment for personality disorders.
  Sessions program:
  * Session 1: Building epistemic trust.
  * Session 2: Introduction to mentalization.
  * Session 3: Mentalization problems.
  * Session 4: Emotions.
  * Session 5: Mentalizing emotions.
  * Session 6: Attachment relationships.
  * Session 7: Attachment and mentalization.
  * Session 8: Interpersonal relationships. Mentalizing relationships in the group.
  * Session 9: Anxiety, attachment and mentalization.
  * Session 10: Depression, attachment and mentalization.
  * Session 11: Flexible content depending on pending topics or participants' needs. Preparing for closing
  * Session 12: Final balance and closing.
  Arms: Brief mentalization-based group psychotherapy
Behavioral: Acceptance and Commitment Therapy group intervention — The intervention includes 12 sessions based on Acceptance and Commitment Therapy. Sessions program:
  * Session 1: Presentation.
  * Session 2: Cognitive defusion
  * Session 3: Uncontrollability of thought, emotions and behavior.
  * Session 4: Creative Hopelessness.
  * Session 5: Mindfulness and acceptance.
  * Session 6: Values.
  * Session 7: Values and action.
  * Session 8: Vital goals.
  * Session 9: Goal achievement plan.
  * Session 10: Implementation.
  * Session 11: Flexible content depending on pending topics or participants' needs. Preparing for closing
  * Session 12: Final balance and closing.
  Arms: Acceptance and commitment therapy group intervention

SUMMARY:
This randomized clinical trial aims to evaluate the effects of mentalization-based group psychotherapy in patients diagnosed with anxiety and/or depression disorders. In total 100 users of mental health communitary services will be recruited for this study. Participants will be randomized in two parallel groups: to receive usual acceptance and commitment therapy group intervention (control group) or to receive brief mentalization-based group psychotherapy (intervention group). Participants in the trial will be assessed at baseline and at 3 months.

DETAILED DESCRIPTION:
QUALITY ASSURANCE PLAN. The researchers will review and report the process during the trial covering participant enrolment, consent and eligibility to protect participants, including reporting of harm and completeness, accuracy and timeliness of data collection.

STANDARD OPERATING PROCEDURES. Participants will be identified from community mental health services who meet all the study eligibility criteria (listed in section Eligibility). Participants will be recruited over a period of 20 months by mental health professionals (clinical psychology residents). Community sample for validation will be recruited by social media. Participants will not receive financial reimbursement for taking part in this trial.

DATA DICTIONARY. All variables collected in this study are listed and described in an electronic case report form, with associated guidelines, to ensure consistency in all gathered data. The following data will be collected in this trial:

Sociodemographical data. Anxiety symptoms: Generalized Anxiety Disorder 7-item scale (GAD-7) Depressice symptoms: Patient Health Questionnaire-9 (PHQ-9) Epistemic Trust: The Epistemic Trust Questionnaire (QET) Epistemic Trust, Mistrust and Credulity: The Epistemic Trust, Mistrust and Credulity Questionnaire (ETMCQ).

Reflective functioning: The Reflective Functioning Questionnaire (RFQ-8) Functional impact: The Work and Social Adjustment Scale (WSAS) Satisfaction with therapy: The Consumer Reports Effectiveness Score (CRES-4)

SAMPLE SIZE ASSESSMENT. The study has sensitivity to detect effect sizes that are considered clinically significant (Cohen's d =0.50) for a power of 0.8, an Alpha of 0.05 and an estimated sample of 100 participants. The calculation was performed with the GPower 3.1.9.2 program for a mean difference with a t-test for two independent groups.

For the validation of the QET, taking into account the subject-item ratio of at least 5: 1 (24 items), and considering the minimum number of recommended subjects to perform an Exploratory Factor Analysis, the minimum number of participants must be 150.Thus, estimating losses of 20%, the total number of participants estimated for the validation is n = 180 .

STATISTICS ANALYSIS PLAN. The analysis will be made following an intention-to-treat procedure. The change of means in the primary outcome variable between the two study groups will be analyzed with the Student's t-test for independent samples if the criteria for its application are met. If the criteria for its application are not met, nonparametric tests will be used. For continuous secondary variables, this test will also be used. A multivariate analysis of variance (ANCOVA) will also be considered to introduce any possible covariate that differs between the two comparison groups in the first evaluation. Potential confounding variables will include gender, age, previous level of depression and anxiety, and diagnosis. A 95% confidence level will be used for all comparisons. The R program will be used for all statistical analyses.

PLAN FOR MISSING DATA. Each researcher is responsible for ensuring that any missing data will be reported as missing in the study database. Procedures can sometimes be considered when using statistical methods that fail in the presence of any missing values, or when in the case of multiple-predictor statistical models all the data for an individual would be omitted because of a missing value in one of the predictors. For analyses involving multiple regression analysis, a multiple imputation approach will be considered and used if statistically sound, depending on the proportion and pattern of missing values.

METHODS TO ENSURE VALIDITY AND QUALITY OF DATA. Accurate and reliable data collection will be assured by verification and cross-check of the case report form (CRF) against the researcher´s records (source document verification). Source document verification will be conducted for 5% of data in subjects. Discrepancies and queries will be generated accordingly in the CRF for online resolution by the researcher at the site. In addition, the CRF data will be reviewed on an ongoing basis for medical and scientific plausibility.

ELIGIBILITY:
Inclusion Criteria:

* Participants are 18 years or older.
* Participants have a diagnosis of ICD-10 F32, F33, F34, F41.1, F41.2, F43 or F43.2.
* Participants have minimal relational skills to participate in group therapy.
* Participants agree to be part of the study by giving signed written consent.

Exclusion Criteria:

* Participants have a diagnosis of ICD-10 F10-19, F20-29, F31, F42, F43.1, F60.
* Participants with cognitive deficits assessed during the initial interview or diagnosis of ICD-10 F70-79.
* Participants with planning or structured suicidal ideation.
* Participants with difficulties in relational skills evaluated during the initial interview.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2024-04-28 (Actual); Primary Completion 2026-05-29 (Estimated); Study Completion 2026-06 (Estimated)

PRIMARY OUTCOMES:
Change from baseline anxiety symptoms at 3 months. | At baseline then at 3 months.
  Generalized Anxiety Disorder 7-item scale (GAD-7), is a self-report questionnaire used to assess the severity of generalized anxiety disorder symptoms. It consists of seven questions that ask respondents to rate how often they have experienced various anxiety-related symptoms over the past two weeks. Each item is scored from 0 (not at all) to 3 (nearly every day), allowing for a total score ranging from 0 to 21. Higher scores indicate greater anxiety severity. The Spanish adaptation used in this study has excellent psychometric properties, with a Cronbach's alpha of .94
Change from baseline depressive symptoms at 3 months. | At baseline then at 3 months.
  Patient Health Questionnaire-9 (PHQ-9) is a self-report tool designed to assess the severity of depression symptoms. It consists of 9 questions using a Lykert-type scale from 0 (not at all) to 3 (nearly every day). Respondents are asked to rate how often they have experienced specific symptoms over the past two weeks. The total score can range from 0 to 27, with higher scores indicating more severe depressive symptoms.

SECONDARY OUTCOMES:
Change from baseline epistemic trust at 3 months. | At baseline then at 3 months.
  The Epistemic Trust Questionnaire (QET) is a 24-item self-report scale to assess the clinical characteristics of Epistemic Trust. The items, rated on a 5-point Likert-type scale scale, cover areas related to hypervigilance, curiosity, and expectancy and openness to help. The original English version show adequate validity and reliability in clinical populations with personality disorder diagnoses and non-clinical populations.
Change from baseline epistemic trust, Mistrust and Credulity at 3 months | At baseline then at 3 months.
  The Epistemic Trust, Mistrust, and Credulity Questionnaire (ETMCQ) is a15-items self-report measure to assess various forms of epistemic stance. The ETMCQ consists of three subscales, namely trust, mistrust, and credulity. Responses were rated across a 7-point Likert scale ranging from "strongly disagree" (= 1) to "strongly agree" (= 7). The questionnaire also showed good reliability and validity.
Change from baseline reflective functioning at 3 months. | At baseline then at 3 months.
  The Reflective Functioning Questionnaire (RFQ-8) is an eight-item self-report instrument to evaluate mentalization. It asks subjects to express their agreement with each item on a 7-point Likert scale (ranging from 1 = "completely disagree" to 7 = "completely agree"). Higher levels of uncertainty regarding mental states were found to be correlated with difficulties in affect regulation, symptoms of psychopathology, interpersonal problems, and attachment anxiety. The spanish validation of the RFQ shows an adequate reliability and validity assessing failures in reflective functioning in general population and personality disorders.
Change from baseline functional impact at 3 months. | At baseline then at 3 months.
  The Work and Social Adjustment Scale (WSAS) is a 5-item self-report scale on functional impairment attributable to an identified mental health problem. The items cover areas related to work, home, social leisure, personal leisure and interpersonal relationships. The Spanish validation confirm the validity and reliability of the scale.
Satisfaction with therapy | At 3 months
  The Consumer Reports Effectiveness Score (CRES-4) consists of 4 items: a satisfaction question, a question to rate the degree of resolution of the main problem, a question about the emotional state before starting treatment and, finally, a question about the emotional state at the time of answering the CRES-4. From these 4 questions, three components can be extracted that correspond to the perception of change in emotional state, satisfaction and problem solving.

CONTACTS AND LOCATIONS:
Locations (1):
- Instituto de Investigacion Biomedica de Malaga - IBIMA, Málaga, Malaga, Spain

REFERENCES:
- [Background] Luyten P, Campbell C, Allison E, Fonagy P. The Mentalizing Approach to Psychopathology: State of the Art and Future Directions. Annu Rev Clin Psychol. 2020 May 7;16:297-325. doi: 10.1146/annurev-clinpsy-071919-015355. Epub 2020 Feb 5. PMID 32023093
- [Background] Fonagy P, Luyten P, Allison E, Campbell C. Mentalizing, Epistemic Trust and the Phenomenology of Psychotherapy. Psychopathology. 2019;52(2):94-103. doi: 10.1159/000501526. Epub 2019 Jul 30. PMID 31362289
- [Background] Campbell C, Tanzer M, Saunders R, Booker T, Allison E, Li E, O'Dowda C, Luyten P, Fonagy P. Development and validation of a self-report measure of epistemic trust. PLoS One. 2021 Apr 16;16(4):e0250264. doi: 10.1371/journal.pone.0250264. eCollection 2021. PMID 33861805
- [Background] Ruiz-Parra E, Manzano-Garcia G, Mediavilla R, Rodriguez-Vega B, Lahera G, Moreno-Perez AI, Torres-Cantero AM, Rodado-Martinez J, Bilbao A, Gonzalez-Torres MA. The Spanish version of the reflective functioning questionnaire: Validity data in the general population and individuals with personality disorders. PLoS One. 2023 Apr 6;18(4):e0274378. doi: 10.1371/journal.pone.0274378. eCollection 2023. PMID 37023214
- [Background] Kroenke K, Spitzer RL, Williams JB. The PHQ-9: validity of a brief depression severity measure. J Gen Intern Med. 2001 Sep;16(9):606-13. doi: 10.1046/j.1525-1497.2001.016009606.x. PMID 11556941
- [Background] Spitzer RL, Kroenke K, Williams JB, Lowe B. A brief measure for assessing generalized anxiety disorder: the GAD-7. Arch Intern Med. 2006 May 22;166(10):1092-7. doi: 10.1001/archinte.166.10.1092. PMID 16717171
- [Background] Mundt JC, Marks IM, Shear MK, Greist JH. The Work and Social Adjustment Scale: a simple measure of impairment in functioning. Br J Psychiatry. 2002 May;180:461-4. doi: 10.1192/bjp.180.5.461. PMID 11983645
- [Background] Knapen S, Swildens WE, Mensink W, Hoogendoorn A, Hutsebaut J, Beekman ATF. The development and psychometric evaluation of the Questionnaire Epistemic Trust (QET): A self-report assessment of epistemic trust. Clin Psychol Psychother. 2023 Nov 10. doi: 10.1002/cpp.2930. Online ahead of print. PMID 37947067